CLINICAL TRIAL: NCT06086015
Title: Non-invasive Neuromodulation of the Right Anterior Amygdala Using tACS: A Double-blind Randomized Sham Controlled Clinical Trial for the Treatment of Anxiety Related Disorders With an Open-Label Extension
Brief Title: Apply tACS to Alleviate Anxiety Symptoms
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: NeuroCognitive and Behavioral Institute Clinical Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AMG-05
Record Dates: First submitted 2023-10-05; First posted 2023-10-17 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Anxiety Disorders
MeSH Terms: conditions — Anxiety Disorders | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active group (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS)
- Sham group (Placebo Comparator)
  Interventions: Device: transcranial alternating current stimulation (tACS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — 2mA tACS over right hemisphere, at positions F4, P4, T8 (10-10 convention)

SUMMARY:
This is a clinical research trial exploring the efficacy of non-invasive neuromodulation (NM) intervention in the treatment of anxiety. The NM used in this study consists of 25 minutes of 5 hz transcranial alternating current stimulation (tACS) titrated up to 2mA targeting the anterolateral amygdala across 12 treatment sessions with a 3-4 week time period. The studied population includes patients with the following anxiety disorders: generalized anxiety disorder (GAD), social anxiety disorder (SAD), separation anxiety disorder of childhood, and post-traumatic stress disorder (PTSD). Participants will be randomly assigned to tACS or sham, cross-over, then followed by an optional open-label extension phase.

ELIGIBILITY:
Inclusion Criteria:

* Meet SCID-5/MINI KID criteria for one of the above-mentioned anxiety disorders.
* Subject, or legally acceptable representative (LAR), is able to read, understand, and provide written informed consent and assent, as applicable.
* Subjects requiring an LAR will have an identified caregiver who meets the following criteria: Able to reliably report and communicate on the subject's level of functioning and either lives with the subject or sees the subject on average for ≥ 3 hours/day ≥ 4 days/week, or receives reports from a caregiver, such as an aide, who meets this criteria, and in the investigator's opinion - the extent of contact is sufficient to provide meaningful assessment of changes in subject behavior and function over time
* Able to be compliant with all study procedures
* Age range: 5 years of age or older
* Stable medications for non-excluded concurrent medical conditions for eight weeks prior to randomization
* If receiving psychotherapy, participants must have started psychotherapy at least 2 months prior to randomization
* Health: Physically acceptable for the study with no expected medical conditions likely to occur during or immediately after the study, as confirmed by medical history
* Clinical laboratory values of TSH and T4, within 90 days from randomization must be within normal limits or judged not clinically related by the physician sub-investigator or PI to the subject's cognitive impairment if abnormalities are present.

Exclusion Criteria:

1. Neurodegenerative disease
2. Epilepsy
3. Intellectual Disability
4. Pregnancy or lactation
5. Convexity skull defects
6. Raised intracranial pressure
7. Intracranial electrodes
8. Vascular clips or shunts in the brain
9. Cardiac pacemakers or other implanted biomedical devices
10. An active medical disorder that could explain, in the opinion of the PI or by medical history, the anxiety disorder.
11. Had an abrupt and significant change in functioning within 3 months of randomization.
12. Meets criteria for any substance use addiction as defined by DSM-5/SCID-5 CV.
13. Active alcoholism as defined by 3 or more bottles of beer or glasses of wine or 2 hard liquor drinks per day/night 3 or > times per week at any time within the past 12 weeks of screening or any other addiction to non-prescription substances.
14. Schizophrenia spectrum disorders and bipolar spectrum disorders.
15. Active suicidal tendency (evaluated by Columbia-Suicide Severity Rating Scale [C-SSRS], traditional version). Note: If the BDI or CDS of the participants significantly increase, the CSSRS will be repeated.
16. Unstable medical condition (including expected medication change/titration).
17. Premenstrual dysphoric disorder.
18. Factious/malingering disorder and any patients applying for disability warranty.
19. Somatoform disorders subtypes: conversion and hypochondriasis.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate informed by Beck Anxiety Inventory (BAI) | 12 treatment sessions, with 3-4 sessions/week, and the time frame for each participant is 3 to 4 weeks.
  BAI is a self-rated scale, with scores ranging from 0 to 63. We will calculate the treatment response rate as (pre-treatment BAI minus post-treatment BAI)/pre-treatment BAI
Hamilton Anxiety Rating Scale (HAMA) | 12 treatment sessions, with 3-4 sessions/week, and the time frame for each participant is 3 to 4 weeks.
  HAMA is a clinician-rated scale, with scores ranging from 0 to 56. We will calculate the treatment response rate as (pre-treatment HAMA minus post-treatment HAMA)/pre-treatment HAMA. We will compute the average of response rates from HAMA and BAI as the final outcome measure.

SECONDARY OUTCOMES:
PTSD Checklist (PCL) for PTSD cohort | 12 treatment sessions, with 3-4 sessions/week, and the time frame for each participant is 3 to 4 weeks.
  For the PTSD patients, in addition to anxiety measurement, we will also use PCL (ranges from 0 to 80) to register the symptom severity change. Again, the outcome measure is the treatment response rate, defined as pre-treatment PCL minus post-treatment PCL)/pre-treatment PCL

CONTACTS AND LOCATIONS:
Overall Officials: Gerald Tramontano, Principal Investigator — NCI Clinical Research Foundation
Locations (1):
- NCI Clinical Research Foundation, Mount Arlington, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No